CLINICAL TRIAL: NCT00375440
Title: Randomized Placebo Controlled Study Using Tranexamic Acid in Revision Total Hip Arthroplasty
Brief Title: Tranexamic Acid Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely as investigator left the institution.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Alexander Rosenstein, MD
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: L05-063
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Tranexamic Acid; Revision Total Hip Replacement; Reduction in Blood Loss
MeSH Terms: interventions — Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid

SUMMARY:
The purpose of this study is to determine if tranexamic acid significantly reduces blood loss and blood transfusion in revision total hip replacement. Tranexamic acid is a drug that helps to reduce blood loss during surgery. Revision total hip replacement surgery is treatment for patients who have previously had hipe replacement surgery which failed and must be repaired/replaced.

DETAILED DESCRIPTION:
Tranexamic acid is an anti-fibrinolytic agent that inhibits fibrinolysis leading to a reduction of blood loss without concurrently increasing the risk of thromboembolic complications. Several studies have shown that tranexamic acid reduces blood loss and blood transfusions in primary total hip and knee arthroplasty. However, there have not been any studies that evaluate its efficacy in revision total hip arthroplasty. The significance of this study is that the need for blood transfusions and their complications may be minimized in revision hip arthroplasty if tranexamic acid is found to significantly decrease the amount of blood transfusions.

After the patient has been consented, he or she will be randomized into one of two groups (tranexamic acid and placebo) by the School of Pharmacy. The placebo will be crystalloid fluid of equal volume as tranexamic acid. The patient will then undergo revision total hip arthroplasty by Dr. Rosenstein and be administered tranexamic acid or placebo. Blood loss will be recorded intraoperatively and postoperatively through drains. Criteria for blood transfusion include hemoglobin less than 10g/dl or hematocrit less than 30%. Once the operation ends, the drug or placebo will be discontinued and the postoperative care is unchanged from current standards/protocols. Intraoperative blood loss, total blood loss, and number of blood transfusions will be recorded and analyzed. Length of acute hospital stay will also be recorded. A cost analysis will be performed comparing tranexamic acid to blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Failed primary total hip arthroplasty (femoral stem, acetabular component, or both)
* 18-100 years of age

Exclusion Criteria:

* Prosthetic infection
* Primary total hip arthroplasty
* Prisoners
* Pregnancy
* Previous adverse reaction to tranexamic acid
* Bleeding/coagulation disorders
* Renal insufficiency (serum creatinine>two standard deviations for age)
* History of deep venous thrombosis or pulmonary embolism
* Religious beliefs/practices prohibiting blood transfusions
* Wards of the state
* Cognitively impaired patients
* Terminally ill patients
* Students and/or employees
* Color blindness

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Introperative blood loss
Total blood loss
Number of blood transfusions required

SECONDARY OUTCOMES:
Length of acute hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Alexander D Rosenstein, MD, Principal Investigator — Texas Tech University Health Sciences Center Department of Orthopaedic Surgery
Locations (1):
- Texas Tech University Health Sciences Center Department of Orthopaedic Surgery, Lubbock, Texas, United States

REFERENCES:
- [Background] Benoni G, Lethagen S, Nilsson P, Fredin H. Tranexamic acid, given at the end of the operation, does not reduce postoperative blood loss in hip arthroplasty. Acta Orthop Scand. 2000 Jun;71(3):250-4. doi: 10.1080/000164700317411834. PMID 10919295
- [Background] Benoni G, Fredin H, Knebel R, Nilsson P. Blood conservation with tranexamic acid in total hip arthroplasty: a randomized, double-blind study in 40 primary operations. Acta Orthop Scand. 2001 Oct;72(5):442-8. doi: 10.1080/000164701753532754. PMID 11728069
- [Background] D'Ambrosio A, Borghi B, Damato A, D'Amato G, Antonacci D, Valeri F. Reducing perioperative blood loss in patients undergoing total hip arthroplasty. Int J Artif Organs. 1999 Jan;22(1):47-51. PMID 10098585
- [Background] Ekback G, Axelsson K, Ryttberg L, Edlund B, Kjellberg J, Weckstrom J, Carlsson O, Schott U. Tranexamic acid reduces blood loss in total hip replacement surgery. Anesth Analg. 2000 Nov;91(5):1124-30. doi: 10.1097/00000539-200011000-00014. PMID 11049894
- [Background] Garneti N, Field J. Bone bleeding during total hip arthroplasty after administration of tranexamic acid. J Arthroplasty. 2004 Jun;19(4):488-92. doi: 10.1016/j.arth.2003.12.073. PMID 15188109
- [Background] Hayes A, Murphy DB, McCarroll M. The efficacy of single-dose aprotinin 2 million KIU in reducing blood loss and its impact on the incidence of deep venous thrombosis in patients undergoing total hip replacement surgery. J Clin Anesth. 1996 Aug;8(5):357-60. doi: 10.1016/0952-8180(96)00080-3. PMID 8832445
- [Background] Hiippala ST, Strid LJ, Wennerstrand MI, Arvela JV, Niemela HM, Mantyla SK, Kuisma RP, Ylinen JE. Tranexamic acid radically decreases blood loss and transfusions associated with total knee arthroplasty. Anesth Analg. 1997 Apr;84(4):839-44. doi: 10.1097/00000539-199704000-00026. PMID 9085968
- [Background] Ho KM, Ismail H. Use of intravenous tranexamic acid to reduce allogeneic blood transfusion in total hip and knee arthroplasty: a meta-analysis. Anaesth Intensive Care. 2003 Oct;31(5):529-37. doi: 10.1177/0310057X0303100507. PMID 14601276
- [Background] Husted H, Blond L, Sonne-Holm S, Holm G, Jacobsen TW, Gebuhr P. Tranexamic acid reduces blood loss and blood transfusions in primary total hip arthroplasty: a prospective randomized double-blind study in 40 patients. Acta Orthop Scand. 2003 Dec;74(6):665-9. doi: 10.1080/00016470310018171. PMID 14763696
- [Background] Ido K, Neo M, Asada Y, Kondo K, Morita T, Sakamoto T, Hayashi R, Kuriyama S. Reduction of blood loss using tranexamic acid in total knee and hip arthroplasties. Arch Orthop Trauma Surg. 2000;120(9):518-20. doi: 10.1007/s004029900132. PMID 11011672
- [Background] Janssens M, Joris J, David JL, Lemaire R, Lamy M. High-dose aprotinin reduces blood loss in patients undergoing total hip replacement surgery. Anesthesiology. 1994 Jan;80(1):23-9. doi: 10.1097/00000542-199401000-00007. PMID 7507304
- [Background] Jeserschek R, Clar H, Aigner C, Rehak P, Primus B, Windhager R. Reduction of blood loss using high-dose aprotinin in major orthopaedic surgery: a prospective, double-blind, randomised and placebo-controlled study. J Bone Joint Surg Br. 2003 Mar;85(2):174-7. doi: 10.1302/0301-620x.85b2.13303. PMID 12678347
- [Background] Kasper SM, Elsner F, Hilgers D, Grond S, Rutt J. A retrospective study of the effects of small-dose aprotinin on blood loss and transfusion needs during total hip arthroplasty. Eur J Anaesthesiol. 1998 Nov;15(6):669-75. doi: 10.1097/00003643-199811000-00008. PMID 9884852
- [Background] Langdown AJ, Field J, Grote J, Himayat H. Aprotinin (Trasylol) does not reduce bleeding in primary total hip arthroplasty. J Arthroplasty. 2000 Dec;15(8):1009-12. doi: 10.1054/arth.2000.8102. PMID 11112196
- [Background] Lemay E, Guay J, Cote C, Roy A. Tranexamic acid reduces the need for allogenic red blood cell transfusions in patients undergoing total hip replacement. Can J Anaesth. 2004 Jan;51(1):31-7. doi: 10.1007/BF03018543. PMID 14709457
- [Background] Murkin JM, Shannon NA, Bourne RB, Rorabeck CH, Cruickshank M, Wyile G. Aprotinin decreases blood loss in patients undergoing revision or bilateral total hip arthroplasty. Anesth Analg. 1995 Feb;80(2):343-8. doi: 10.1097/00000539-199502000-00023. PMID 7529467
- [Background] Murkin JM, Haig GM, Beer KJ, Cicutti N, McCutchen J, Comunale ME, Hall R, Ruzicka BB. Aprotinin decreases exposure to allogeneic blood during primary unilateral total hip replacement. J Bone Joint Surg Am. 2000 May;82(5):675-84. doi: 10.2106/00004623-200005000-00008. PMID 10819278
- [Background] Tanaka N, Sakahashi H, Sato E, Hirose K, Ishima T, Ishii S. Timing of the administration of tranexamic acid for maximum reduction in blood loss in arthroplasty of the knee. J Bone Joint Surg Br. 2001 Jul;83(5):702-5. doi: 10.1302/0301-620x.83b5.11745. PMID 11476309
- [Background] Walsh TS, McClelland DB. When should we transfuse critically ill and perioperative patients with known coronary artery disease? Br J Anaesth. 2003 Jun;90(6):719-22. doi: 10.1093/bja/aeg109. No abstract available. PMID 12765883
- [Background] Yamasaki S, Masuhara K, Fuji T. Tranexamic acid reduces blood loss after cementless total hip arthroplasty-prospective randomized study in 40 cases. Int Orthop. 2004 Apr;28(2):69-73. doi: 10.1007/s00264-003-0511-4. Epub 2003 Oct 10. PMID 15224162